CLINICAL TRIAL: NCT06708442
Title: Guided Narrative Technique After Coronavirus Outbreak Influencing Positive and Negative Emotions and Cognition for Children--A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Hubei primary school RCT
Record Dates: First submitted 2024-11-24; First posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Anxiety and Depression
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Writing Group A (WA) (Experimental): First, the guardian of the participant will read the informed consent. After the guardian signs the informed consent, the participant will complete the demographic, emotional and cognitive pre-assessment. The participant will then receive a group cognitive behavioral intervention for 40 minutes each day in the following 3 days. The intervention will take place in school classrooms in a format similar to offline school classes. The therapists are one senior undergraduate and one first-year PhD student from the School of Psychological and Cognitive Sciences who have received sufficient training. The intervention based on the theory of children's cognitive behavioral therapy, with a self-compiled manual. The three sessions are aimed at emotional awareness and management, thoughts recognition, and coping. Each session will be accompanied by the presence of the head teachers.
  Interventions: Behavioral: School-based CBT intervention; Behavioral: Guided Narrative Technique (GNT) Writing
- Drawing Group A (DA) (Active Comparator): For DA group, the procedures of informed consent, pre assessments, cognitive behavior group intervention, and follow-up assessments will be the same as those for WA. After completing the group intervention, the participants in DA will be required to complete the GNT drawing in accordance with the guidelines at a fixed time each day, under the guidance and supervision of the school teachers, and to complete two short mood tests and the post-painting assessments in the following 3 days. Each drawing session will last for 20-30 minutes.
  Interventions: Behavioral: School-based CBT intervention; Behavioral: Guided Narrative Technique (GNT) drawing

INTERVENTIONS:
Behavioral: School-based CBT intervention — School-based CBT intervention: a 3-day, 40-minute per day cognitive behavioral intervention. The intervention will take place in a school classroom in a format similar to offline classroom lectures and classroom interactions. The intervention will lead by one undergraduate student from the School of Psychological and Cognitive Sciences and one first-year doctoral student with training in clinical psychology. The content of the intervention was based on the theory of cognitive behavioral therapy for children, with a complete self-developed intervention manual, and three interventions targeting emotional awareness and management, thought recognition, and problem coping, respectively.
Behavioral: Guided Narrative Technique (GNT) Writing — Guided Narrative Technique (GNT) Writing : GNT writing is an intervention through writing. It will be conducted once a day for 20-30 minutes for three days. Subjects will be asked to complete Guided Narrative Writing at a set time each day for three consecutive days, under the guidance and supervision of a school teacher, following guidelines.
  Arms: Intervention Writing Group A (WA)
Behavioral: Guided Narrative Technique (GNT) drawing — Guided Narrative Technique (GNT) Drawing: GNT drawing is an intervention through drawing. It will be conducted once a day for 20-30 minutes for three days. Subjects will be asked to complete Guided Narrative Drawing at a set time each day for three consecutive days, under the guidance and supervision of a school teacher, following guidelines.
  Arms: Drawing Group A (DA)

SUMMARY:
At the beginning of 2020, the COVID-19 broke out in Wuhan, raging across the country quickly afterwards. As a sudden public health emergency, this epidemic caused some stress reactions (including emotional, cognitive, and behavioral reactions) in children. These stress responses, in moderation, may be beneficial as a response to the challenge. However, excessive, and inappropriate stress responses may damage children's mental health, immune function, and daily function.

School-based CBT intervention is effective in alleviating children and adolescent anxiety. However, the effect last only shortly. Therefore, adding a new intervention component is necessary. Guided Narrative Technique (GNT) is an intervention focusing on narrative coherence and emotional expression. It has writing and drawing versions. The writing version was developed from Expressive Writing and has a significant effect on the improvement of various negative emotions and negative cognitions of traumatized individuals.

In this study, a randomized controlled experiment will be implemented. All participants will take a CBT course first. Then, they will be asked to write or draw about the epidemic or other life events using GNT. The study will explore the impact of CBT course combined with GNT on negative emotions and cognition of children after such a public crisis.

ELIGIBILITY:
Inclusion Criteria:

* have the ability to read and write in Chinese

Exclusion Criteria:

* no parental consent

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 220 (Actual)
Dates: Start 2020-12-02 (Actual); Primary Completion 2021-06-11 (Actual); Study Completion 2021-06-11 (Actual)

PRIMARY OUTCOMES:
Anxiety and depression | From enrollment to the 6-month follow-up
  Child anxiety and depression symptoms measured by RCADS-25.

SECONDARY OUTCOMES:
PTSD for children | From enrollment to the 6-month follow-up
  The Child PTSD Symptom Scale for DSM-5 (CPSS-5) for adolescents and children (scores from 0 to 4, and total scores vary from 0 to 80). A higher score represents worse PTSD symptoms.

OTHER OUTCOMES:
Emotion awareness | From enrollment to the 6-month follow-up
  A 30-item Emotion awareness questionnaire measures emotion awareness on a 3-point Likert scale (1 to 3, and total scores vary from 30 to 90). A higher score represents better emotion awareness.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University, Beijing, China

IPD SHARING:
Plan to Share IPD: No